CLINICAL TRIAL: NCT01360645
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial of the Safety and Efficacy of Fixed Dose OPC-34712 as Adjunctive Therapy in the Treatment of Adults With Major Depressive Disorder, the Pyxis Trial
Brief Title: Study of the Safety and Efficacy of Fixed Dose OPC-34712 as Adjunctive Therapy in the Treatment of Adults With Major Depressive Disorder (the Pyxis Trial)
Acronym: Pyxis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 331-10-228
Record Dates: First submitted 2011-05-24; First posted 2011-05-25 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-10

CONDITIONS: Depressive Disorder; Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders
Keywords: OPC-34712; brexpiprazole; Major Depressive Disorder; Adjunctive Treatment
MeSH Terms: conditions — Depressive Disorder; Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders | interventions — Androgen Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase B (Experimental): Drug: OPC-34712 + ADT
  Drug: Placebo + ADT
  Interventions: Drug: OPC-34712 + ADT; Drug: Placebo + ADT
- Phase A (Placebo Comparator): Intervention: Drug: Placebo + ADT
  Interventions: Drug: Placebo + ADT

INTERVENTIONS:
Drug: OPC-34712 + ADT — Tablet, Oral, 2 mg OPC-34712 and FDA Approved Antidepressant Therapy (ADT)
  Arms: Phase B
Drug: Placebo + ADT — Placebo + FDA Approved Antidepressant (ADT)
  Arms: Phase B
Drug: Placebo + ADT — Placebo + FDA Approved Antidepressant (ADT)
  Arms: Phase A

SUMMARY:
To compare the effect of OPC-34712 (brexpiprazole) to the effect of placebo (an inactive substance) as add on treatment to an assigned FDA approved antidepressant treatment (ADT) in patients with Major Depressive Disorder who demonstrate an incomplete response to a prospective trial of the same assigned FDA approved ADT

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 65 years of age, with diagnosis of major depressive disorder, as defined by DSM-IV-TR criteria
* The current depressive episode must be equal to or greater than 8 weeks in duration
* Subjects must report a history for the current depressive episode of an inadequate response to no more than three adequate antidepressant treatments

Exclusion Criteria:

* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving study drug
* Subjects who report an inadequate response to more than three adequate trials of antidepressant treatments during current depressive episode at a therapeutic dose for an adequate duration.
* Subjects with a current Axis I (DSM-IV-TR) diagnosis of: Delirium, dementia, amnestic or other cognitive disorder, Schizophrenia, schizoaffective disorder, or other psychotic disorder, Bipolar I or II disorder
* Subjects with a clinically significant current Axis II (DSM-IV-TR) diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal or histrionic personality disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 826 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (57):
- United States (37):
  - Research Site, Arcadia, California
  - Research Site, Beverly Hills, California
  - Research Site, Fresno, California
  - Research Site, Oceanside, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Sherman Oaks, California
  - Research Site, Denver, Colorado
  - Research Site, Norwalk, Connecticut
  - Research Site, Coral Springs, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Orlando, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Prairie Village, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Belmont, Massachusetts
  - Research Site, Boston, Massachusetts
  - Research Site, Lincoln, Nebraska
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Dayton, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Salem, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Bala-Cynwyd, Pennsylvania
  - Research Site, Bridgeville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, San Antonio, Texas
  - Research Site, Murray, Utah
  - Research Site, Woodstock, Vermont
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
- Canada (3):
  - Research Site, Penticton, British Columbia
  - Research Site, Toronto, Ontario
  - Research Site, Gatineau, Quebec
- France (5):
  - Research Site, Arcachon
  - Research Site, Élancourt
  - Research Site, Orvault
  - Research Site, Palaiseau
  - Research Site, Toulouse
- Poland (8):
  - Research Site, Bełchatów, Poland
  - Research Site, Katowice, Upper Silesia
  - Research Site, Poznan, Woj. Wielkopolskie
  - Research Site, Gdynia
  - Research Site, Kielce
  - Research Site, Lublin
  - Research Site, Tuszyn
  - Research Site, Warsaw
- Slovakia (4):
  - Research Site, Kosice-Barca, Slovakia
  - Research Site, Bratislava
  - Research Site, Levice
  - Research Site, Michalovce

REFERENCES:
- [Derived] Kapadia S, Zhang Z, Ardic F, Patel M, Thase ME, Papakostas GI. Adjunctive brexpiprazole in patients with major depressive disorder who show minimal or partial response to antidepressant treatment: post hoc analysis of randomized controlled trials. Int J Neuropsychopharmacol. 2025 Oct 1;28(10):pyaf074. doi: 10.1093/ijnp/pyaf074. PMID 41055581
- [Derived] Ardic F, Zhang Z, Hogan M. Effects of adjunctive brexpiprazole in patients with major depressive disorder and sleep disturbance: a post hoc analysis of three randomized trials. Front Psychiatry. 2025 Aug 7;16:1618176. doi: 10.3389/fpsyt.2025.1618176. eCollection 2025. PMID 40852147
- [Derived] Kapadia S, Zhang Z, Csoboth C, Patel M, Thase ME, Papakostas GI. Adjunctive brexpiprazole in patients with unresolved symptoms of depression on antidepressant treatment who are early in the disease course: post hoc analysis of randomized controlled trials. Int J Neuropsychopharmacol. 2025 Aug 1;28(8):pyaf050. doi: 10.1093/ijnp/pyaf050. PMID 40607746
- [Derived] McIntyre RS, Bubolic S, Zhang Z, MacKenzie EM, Therrien F, Miguelez M, Boucher M. Effects of Adjunctive Brexpiprazole on Individual Depressive Symptoms and Functioning in Patients With Major Depressive Disorder and Anxious Distress: Post Hoc Analysis of Three Placebo-Controlled Studies. J Clin Psychopharmacol. 2024 Mar-Apr 01;44(2):133-140. doi: 10.1097/JCP.0000000000001825. PMID 38421922
- [Derived] Newcomer JW, Meehan SR, Chen D, Brubaker M, Weiss C. Changes in Metabolic Parameters and Body Weight in Patients With Prediabetes Treated With Adjunctive Brexpiprazole for Major Depressive Disorder: Pooled Analysis of Short- and Long-Term Clinical Studies. J Clin Psychiatry. 2023 Aug 28;84(5):23m14786. doi: 10.4088/JCP.23m14786. PMID 37656180
- [Derived] McIntyre RS, Therrien F, Ismail Z, Meehan SR, Miguelez M, Larsen KG, Chen D, MacKenzie EM, Thase ME. Effects of adjunctive brexpiprazole on patient life engagement in major depressive disorder: Post hoc analysis of Inventory of Depressive Symptomatology Self-Report data. J Psychiatr Res. 2023 Jun;162:71-78. doi: 10.1016/j.jpsychires.2023.04.012. Epub 2023 Apr 12. PMID 37099968
- [Derived] Newcomer JW, Eriksson H, Zhang P, Meehan SR, Weiss C. Changes in Metabolic Parameters and Body Weight in Patients With Major Depressive Disorder Treated With Adjunctive Brexpiprazole: Pooled Analysis of Phase 3 Clinical Studies. J Clin Psychiatry. 2019 Oct 1;80(6):18m12680. doi: 10.4088/JCP.18m12680. PMID 31577867
- [Derived] Hobart M, Zhang P, Weiss C, Meehan SR, Eriksson H. Adjunctive Brexpiprazole and Functioning in Major Depressive Disorder: A Pooled Analysis of Six Randomized Studies Using the Sheehan Disability Scale. Int J Neuropsychopharmacol. 2019 Mar 1;22(3):173-179. doi: 10.1093/ijnp/pyy095. PMID 30508090
- [Derived] McIntyre RS, Weiller E, Zhang P, Weiss C. Brexpiprazole as adjunctive treatment of major depressive disorder with anxious distress: Results from a post-hoc analysis of two randomised controlled trials. J Affect Disord. 2016 Sep 1;201:116-23. doi: 10.1016/j.jad.2016.05.013. Epub 2016 May 12. PMID 27208498
- [Derived] Thase ME, Youakim JM, Skuban A, Hobart M, Augustine C, Zhang P, McQuade RD, Carson WH, Nyilas M, Sanchez R, Eriksson H. Efficacy and safety of adjunctive brexpiprazole 2 mg in major depressive disorder: a phase 3, randomized, placebo-controlled study in patients with inadequate response to antidepressants. J Clin Psychiatry. 2015 Sep;76(9):1224-31. doi: 10.4088/JCP.14m09688. PMID 26301701

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 826 subjects at 59 trial sites in the following 5 countries: United States, Canada, Poland, Slovakia, and France.
Pre-assignment Details: The study consisted of a 7 to 28-day Screening period, an 8-Week single-blind placebo + ADT prospective Phase-A, a 6-Week double-blind randomization Phase-B or single-blind Phase A+ and a Follow-up of 30 (+2) days after the last dose of study medication.
Groups:
- Single-blind Placebo + ADT: In Phase A, participants were administered placebo as an adjunctive therapy to an open label ADT for 8 weeks
- Brexpiprazole 2 mg/Day + ADT: Participants received Brexpiprazole 2 mg/day as an adjunctive therapy over a 2-week period beginning at the Week 8 visit and continued to take the same ADT that was assigned in Phase A at the final dose taken just prior to the Week 8 visit.
- Double-blind Placebo + ADT: Participants received placebo as an adjunctive therapy over a 2-week period beginning at the Week 8 visit and continued to take the same ADT that was assigned in Phase A at the final dose taken just prior to the Week 8 visit.
- Phase A+ Placebo + ADT: Participants who did not meet criteria for randomization and a follow-up of 30 (+2) days after the last dose of study medication were in Phase A+
Period: Placebo+ADT Prospective Phase-A(8 Weeks)
Arm/Group | Single-blind Placebo + ADT | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT | Phase A+ Placebo + ADT
Started | 824 (826 participants were enrolled but 2 participants discontinued trial before taking study medication.) | 0 | 0 | 0
Completed | 710 | 0 | 0 | 0
Not Completed | 114 | 0 | 0 | 0
Not completed — Lost to Follow-up | 16 | 0 | 0 | 0
Not completed — Adverse Event | 19 | 0 | 0 | 0
Not completed — Met Withdrawal Criteria | 16 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 34 | 0 | 0 | 0
Not completed — Protocol Deviation | 24 | 0 | 0 | 0
Not completed — Physician Decision | 5 | 0 | 0 | 0
Period: Phase B (6 Weeks)
Arm/Group | Single-blind Placebo + ADT | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT | Phase A+ Placebo + ADT
Started | 0 | 188 | 191 | 0
Completed | 0 | 174 | 178 | 0
Not Completed | 0 | 14 | 13 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 6 | 0 | 0
Not completed — Met Withdrawal Criteria | 0 | 3 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 8 | 0
Not completed — Protocol Deviation | 0 | 1 | 3 | 0
Period: Phase A+
Arm/Group | Single-blind Placebo + ADT | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT | Phase A+ Placebo + ADT
Started | 0 | 0 | 0 | 331
Completed | 0 | 0 | 0 | 307
Not Completed | 0 | 0 | 0 | 24
Not completed — Lost to Follow-up | 0 | 0 | 0 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Met Withdrawal Criteria | 0 | 0 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5
Not completed — Protocol Deviation | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Randomized sample were used. Randomized sample comprises all who were randomized in Phase B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT | Total
Number analyzed (Participants) | 188 | 191 | 379
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (11.6) | 45.2 (11.3) | 44.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 137 | 267
  Male | 58 | 54 | 112

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (End of Phase A [Week 8]) to Week 14 in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score for the Efficacy Sample.
Description: The MADRS consists of 10 items, all rated on a 0 to 6 scale with 0 being the "best" rating and 6 being the "worst" rating. The MADRS total score is the sum of ratings for all 10 items. The possible total scores are from 0 to 60. The MADRS total score will be un-evaluable if less than 8 of the 10 items are recorded. If 8 or 9 of the 10 items are recorded, the MADRS total score will be the mean of the recorded items multiplied by 10 and then rounded to the first decimal place.
Time Frame: Baseline and Week 14
Population: The Efficacy Sample comprised of all participants in the Safety Sample who had an end of Phase A (i.e, Week 8) value and at least one post-randomization efficacy evaluation for MADRS total score in Phase B.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 187 | 191
Units on a scale | -8.27 (0.61) | -5.15 (0.60)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; The primary analysis was performed on the Efficacy Sample by fitting a Mixed Model Repeated Measures (MMRM) analysis with an unstructured variance covariance structure in which the change from the end of Phase A (Week 8) in MADRS Total Score (at Weeks 9 to 14) was the dependent variable. The model included fixed class effect terms for treatment, trial site, visit week, and an interaction term of treatment by visit week; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -3.12, 95% CI 2-sided [-4.70 to -1.54]

2. Primary Outcome: Change From Baseline (End of Phase A [Week 8]) to Week 14 in MADRS Total Score for the Efficacy Sample Per the Final Protocol.
Description: as for outcome 1
Time Frame: Baseline and Week 14
Population: All participants in the Efficacy Sample who met the revised randomization criteria for incomplete response as defined in Protocol Amendment 3.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 175 | 178
Units on a scale | -8.36 (0.64) | -5.15 (0.63)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -3.21, 95% CI 2-sided [-4.87 to -1.54]

3. Secondary Outcome: Mean Change From Baseline (End of Phase A [Week 8]) to Week 14 in Sheehan Disability Scale (SDS) Score for the Efficacy Sample.
Description: The SDS is a self-rated instrument used to measure the effect of the patient's symptoms on work/school, social life, and family/home responsibilities. For each of the three items, scores range from 0 through 10. The number most representative of how much each area was disrupted by symptoms is marked along the line from 0 = not at all, to 10 = extremely. For the work/school item, no response was to be entered if the patient did not work or go to school for reasons unrelated to the disorder and a response therefore not being applicable. The Mean SDS Score will be calculated over the three item scores. All three item scores need to be available with the exception of the work/school item score when this item is not applicable.
Time Frame: Baseline and Week 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 179 | 181
Units on a scale | -1.35 (0.17) | -0.91 (0.17)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Test type: Superiority or Other; p = 0.0372, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.86 to -0.03]

4. Secondary Outcome: Mean Change From Baseline (End of Phase A [Week 8]) to Week 14 in SDS Score for the Efficacy Sample Per the Final Protocol
Description: as for outcome 3
Time Frame: Baseline and Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 167 | 170
Units on a scale | -1.35 (0.17) | -0.89 (0.17)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Test type: Superiority or Other; p = 0.0349, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.88 to -0.03]

5. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) to Week 14 in MADRS Total Score by Trial Week for the Efficacy Sample.
Description: as for outcome 1
Time Frame: Week 9, 10, 11, 12, and 13
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 187 | 191
Units on a scale
  Week 9 | -3.15 (0.40) | -1.86 (0.39)
  Week 10 | -5.15 (0.47) | -3.43 (0.47)
  Week 11 | -6.69 (0.52) | -4.06 (0.52)
  Week 12 | -7.22 (0.55) | -4.63 (0.54)
  Week 13 | -8.28 (0.58) | -5.10 (0.57)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 9; Test type: Superiority or Other; p = 0.0080, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-2.25 to -0.34]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 10; Test type: Superiority or Other; p = 0.0045, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.72, 95% CI 2-sided [-2.91 to -0.54]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 11; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -2.63, 95% CI 2-sided [-3.96 to -1.30]
Statistical Analysis 4: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 12; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -2.59, 95% CI 2-sided [-4.01 to -1.18]
Statistical Analysis 5: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 13; Test type: Superiority or Other; p = 0.0000, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -3.19, 95% CI 2-sided [-4.68 to -1.70]

6. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) to Week 14 in MADRS Total Score by Trial Week for the Efficacy Sample Per the Final Protocol.
Description: as for outcome 1
Time Frame: Week 9, 10, 11, 12, and 13
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 175 | 178
Units on a scale
  Week 9 | -3.05 (0.41) | -1.74 (0.41)
  Week 10 | -5.04 (0.49) | -3.52 (0.48)
  Week 11 | -6.58 (0.54) | -4.17 (0.53)
  Week 12 | -7.24 (0.58) | -4.72 (0.57)
  Week 13 | -8.28 (0.61) | -5.01 (0.60)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 9; Test type: Superiority or Other; p = 0.0086, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-2.28 to -0.34]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 10; Test type: Superiority or Other; p = 0.0149, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.52, 95% CI 2-sided [-2.74 to -0.30]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 11; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -2.42, 95% CI 2-sided [-3.78 to -1.05]
Statistical Analysis 4: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 12; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -2.52, 95% CI 2-sided [-4.00 to -1.04]
Statistical Analysis 5: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 13; Test type: Superiority or Other; p = 0.0000, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -3.28, 95% CI 2-sided [-4.84 to -3.28]

7. Secondary Outcome: Mean Clinical Global Impression-Improvement (CGI-I) Scale Score (End of Phase A [Week 8]) to Week 14 by Trial Week for the Efficacy Sample.
Description: The items on CGI-I scale are: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse. The score of 0 (= not assessed) will be set to missing. The CGI-I is therefore a 7-point scale from 1 through 7. The CGI-I was measured in related to Baseline (Week 8).
Time Frame: Week 9, 10, 11, 12, 13, and 14
Population: The Efficacy Sample comprised of all participants in the Safety Sample who had an end of Phase A (i.e, Week 8) value and at least one post-randomization efficacy evaluation for MADRS total score in Phase B. The LOCF data set included data recorded at a Phase B visit, if no observation was recorded, data was carried forward from the previous visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 187 | 191
Units on a scale
  Week 9 | 3.41 (0.83) | 3.62 (0.74)
  Week 10 | 3.17 (0.89) | 3.37 (0.82)
  Week 11 | 3.03 (1.02) | 3.23 (0.90)
  Week 12 | 2.84 (0.99) | 3.19 (1.04)
  Week 13 | 2.74 (1.07) | 3.13 (1.06)
  Week 14 | 2.75 (1.13) | 3.13 (1.09)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 9; Test type: Superiority or Other; p = 0.0022, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from Cochran-Mantel-Haenszel (CMH) row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.38 to -0.08]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 10; Test type: Superiority or Other; p = 0.0115, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.38 to -0.05]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 11; Test type: Superiority or Other; p = 0.0255, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.41 to -0.03]
Statistical Analysis 4: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 12; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.57 to -0.16]
Statistical Analysis 5: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 13; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.62 to -0.20]
Statistical Analysis 6: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 14; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.60 to -0.17]

8. Secondary Outcome: Mean CGI-I Scale Score (End of Phase A [Week 8]) to Week 14 by Trial Week for the Efficacy Sample Per the Final Protocol.
Description: as for outcome 7
Time Frame: Week 9, 10, 11, 12, 13, and 14
Population: All participants in the efficacy sample who met the revised randomization criteria for incomplete response as defined in protocol amendment 3. The LOCF data set included data recorded at a Phase B visit, if no observation was recorded, data was carried forward from the previous visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 175 | 178
Units on a scale
  Week 9 | 3.44 (0.81) | 3.67 (0.70)
  Week 10 | 3.21 (0.89) | 3.40 (0.82)
  Week 11 | 3.07 (1.01) | 3.25 (0.89)
  Week 12 | 2.85 (1.01) | 3.23 (1.05)
  Week 13 | 2.78 (1.07) | 3.18 (1.06)
  Week 14 | 2.77 (1.14) | 3.17 (1.10)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 9; Test type: Superiority or Other; p = 0.0010, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.40 to -0.10]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 10; Test type: Superiority or Other; p = 0.0290, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.37 to -0.02]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 11; Test type: Superiority or Other; p = 0.0422, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.40 to -0.01]
Statistical Analysis 4: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 12; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.61 to -0.18]
Statistical Analysis 5: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 13; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.64 to -0.20]
Statistical Analysis 6: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 14; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel; P-value and treatment difference (CI) are derived from CMH row mean score differ test controlling for study center; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.65 to -0.19]

9. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) to Week 14 in Clinical Global Impression - Severity of Illness (CGI-S) Scale Score for the Efficacy Sample.
Description: Items on CGI-S scale are: 0 = not assessed, 1 = normal, not at all ill, 2 = borderline mentally ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill patients. The score 0 (= not assessed) will be set to missing. The CGI-S is therefore a 7-point scale from 1 through 7.
Time Frame: Week 9, 10, 11, 12, 13, and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 187 | 191
Units on a scale
  Week 9 | -0.25 (0.05) | -0.12 (0.05)
  Week 10 | -0.45 (0.05) | -0.31 (0.05)
  Week 11 | -0.61 (0.06) | -0.40 (0.06)
  Week 12 | -0.70 (0.07) | -0.45 (0.06)
  Week 13 | -0.86 (0.07) | -0.50 (0.07)
  Week 14 | -0.91 (0.07) | -0.58 (0.07)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 9; Test type: Superiority or Other; p = 0.0229, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.25 to -0.02]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 10; Test type: Superiority or Other; p = 0.0459, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.28 to -0.00]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 11; Test type: Superiority or Other; p = 0.0097, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.37 to -0.05]
Statistical Analysis 4: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 12; Test type: Superiority or Other; p = 0.0038, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.42 to -0.08]
Statistical Analysis 5: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 13; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.54 to -0.18]
Statistical Analysis 6: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 14; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.52 to -0.15]

10. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) to Week 14 in CGI-S Scale Score for the Efficacy Sample Per the Final Protocol.
Description: as for outcome 9
Time Frame: Week 9, 10, 11, 12, 13, and 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 175 | 178
Units on a scale
  Week 9 | -0.24 (0.05) | -0.09 (0.05)
  Week 10 | -0.43 (0.06) | -0.32 (0.06)
  Week 11 | -0.58 (0.06) | -0.42 (0.06)
  Week 12 | -0.70 (0.07) | -0.46 (0.07)
  Week 13 | -0.85 (0.07) | -0.50 (0.07)
  Week 14 | -0.91 (0.07) | -0.57 (0.07)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 9; Test type: Superiority or Other; p = 0.0109, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.27 to -0.04]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 10; Test type: Superiority or Other; p = 0.1286, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.25 to 0.03]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 11; Test type: Superiority or Other; p = 0.0521, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.32 to 0.00]
Statistical Analysis 4: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 12; Test type: Superiority or Other; p = 0.0084, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.42 to -0.06]
Statistical Analysis 5: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 13; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.54 to -0.16]
Statistical Analysis 6: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 14; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.53 to -0.15]

11. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) to Week 14 in the Inventory of Depressive Symptomatology (Self-Report) (IDS-SR) Total Score for the Efficacy Sample.
Description: The IDS-SR consists of 30 items, all rated on a 0 to 3 scale with 0 being the "best" rating and 3 being the "worst" rating. Besides item 9, two sub-items 9A and 9B exist, with possible scores of 1, 2 or 3 for item 9A, and 0 or 1 for item 9B. The scores for these two sub-items are not included in the calculation of the total score. Item 11 or item 12 should be completed but not both, and similarly, item 13 or item 14 should be completed but not both. Should items 11 and 12 be rated both, then the maximum of the two scores will be used. The same approach will be used for handling items 13 and 14.
  The IDS-SR total score is the sum of ratings of 28 item scores. The possible IDS-SR total score ranges from 0 to 84.
Time Frame: Week 9, 10, 11, 12, 13, and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 187 | 191
Units on a scale
  Week 9 | -3.02 (0.52) | -1.45 (0.51)
  Week 10 | -4.17 (0.59) | -2.64 (0.59)
  Week 11 | -5.41 (0.65) | -4.31 (0.64)
  Week 12 | -6.16 (0.68) | -4.69 (0.67)
  Week 13 | -7.00 (0.72) | -5.25 (0.71)
  Week 14 | -7.49 (0.74) | -5.52 (0.73)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 9; Test type: Superiority or Other; p = 0.0139, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.57, 95% CI 2-sided [-2.82 to -0.32]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 10; Test type: Superiority or Other; p = 0.0436, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-3.01 to -0.04]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 11; Test type: Superiority or Other; p = 0.1903, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-2.75 to 0.55]
Statistical Analysis 4: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 12; Test type: Superiority or Other; p = 0.0951, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.47, 95% CI 2-sided [-3.21 to 0.26]
Statistical Analysis 5: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 13; Test type: Superiority or Other; p = 0.0626, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-3.59 to 0.09]
Statistical Analysis 6: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 14; Test type: Superiority or Other; p = 0.0435, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.96, 95% CI 2-sided [-3.87 to -0.06]

12. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) to Week 14 in the IDS-SR Total Score for the Efficacy Sample Per the Final Protocol.
Description: as for outcome 11
Time Frame: Week 9, 10, 11, 12, 13, and 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 175 | 178
Units on a scale
  Week 9 | -3.30 (0.53) | -1.59 (0.51)
  Week 10 | -4.29 (0.61) | -3.13 (0.60)
  Week 11 | -5.45 (0.67) | -4.73 (0.66)
  Week 12 | -6.32 (0.71) | -5.06 (0.70)
  Week 13 | -7.03 (0.74) | -5.60 (0.73)
  Week 14 | -7.59 (0.77) | -6.05 (0.75)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 9; Test type: Superiority or Other; p = 0.0069, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.71, 95% CI 2-sided [-2.95 to -0.47]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 10; Test type: Superiority or Other; p = 0.1322, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-2.68 to 0.35]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 11; Test type: Superiority or Other; p = 0.4055, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-2.41 to 0.98]
Statistical Analysis 4: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 12; Test type: Superiority or Other; p = 0.1715, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.26, 95% CI 2-sided [-3.08 to 0.55]
Statistical Analysis 5: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 13; Test type: Superiority or Other; p = 0.1424, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.42, 95% CI 2-sided [-3.33 to 0.48]
Statistical Analysis 6: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Week 14; Test type: Superiority or Other; p = 0.1270, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-3.52 to 0.44]

13. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) in SDS Item Scores for the Efficacy Sample.
Description: as for outcome 3
Time Frame: Week 11 and 14
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 187 | 191
Units on a scale
  Item: Work/School: Week 11 | -0.70 (0.21) | -0.42 (0.22)
  Item: Work/School: Week 14 | -1.09 (0.22) | -0.90 (0.22)
  Item: Social life: Week 11 | -1.17 (0.17) | -0.67 (0.17)
  Item: Social life: Week 14 | -1.54 (0.19) | -1.04 (0.18)
  Item: Family life: Week 11 | -1.06 (0.18) | -0.43 (0.18)
  Item: Family life: Week 14 | -1.33 (0.19) | -0.73 (0.19)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; For Item: Work/School: Week 11; Test type: Superiority or Other; p = 0.3079, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.81 to 0.26]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; For Item: Work/School: Week 14; Test type: Superiority or Other; p = 0.4771, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.73 to 0.34]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; For Item: Social life: Week 11; Test type: Superiority or Other; p = 0.0195, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.92 to -0.08]
Statistical Analysis 4: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; For Item: Social life: Week 14; Test type: Superiority or Other; p = 0.0323, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.96 to -0.04]
Statistical Analysis 5: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; For Item: Family life: Week 11; Test type: Superiority or Other; p = 0.0058, Cochran-Mantel-Haenszel; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.07 to -0.18]
Statistical Analysis 6: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; For Item: Family life: Week 14; Test type: Superiority or Other; p = 0.0129, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-1.07 to -0.13]

14. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) in SDS Item Scores for the Efficacy Sample Per the Final Protocol.
Description: as for outcome 3
Time Frame: Week 11 and 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 175 | 178
Units on a scale
  Item: Work/School: Week 11 | -0.76 (0.22) | -0.58 (0.22)
  Item: Work/School: Week 14 | -1.11 (0.23) | -0.96 (0.23)
  Item: Social life: Week 11 | -1.18 (0.18) | -0.69 (0.18)
  Item: Social life: Week 14 | -1.57 (0.19) | -1.02 (0.19)
  Item: Family life: Week 11 | -0.99 (0.19) | -0.43 (0.18)
  Item: Family life: Week 14 | -0.43 (0.18) | -0.70 (0.19)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Item: Work/School Week 11; Test type: Superiority or Other; p = 0.5151, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.71 to 0.36]
Statistical Analysis 2: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Item: Work/School Week 14; Test type: Superiority or Other; p = 0.6080, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.70 to 0.41]
Statistical Analysis 3: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Item: Social life-Week 11; Test type: Superiority or Other; p = 0.0267, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.92 to -0.06]
Statistical Analysis 4: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Item: Social life-Week 14; Test type: Superiority or Other; p = 0.0224, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-1.01 to -0.08]
Statistical Analysis 5: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Item: Family life-Week 11; Test type: Superiority or Other; p = 0.0146, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-1.01 to -0.11]
Statistical Analysis 6: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Statistical analysis for Item: Family life-Week 14; Test type: Superiority or Other; p = 0.0113, Mixed Models Analysis; MMRM method was used with trial site; treatment group-visit; Baseline-visit interaction as an unstructured covariate; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.09 to -0.14]

15. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) to Week 14 in Hamilton Depression (HAM-D) Rating Scale Total Score for the Efficacy Sample.
Description: The HAM-D (17-Item) consists of 17 items. Eight items are rated on a 0 to 2 scale (items 4, 5, 6, 12, 13, 14, 16 and 17), while nine items (items 1, 2, 3, 7, 8, 9, 10, 11, and 15) are rated on a 0 to 4 scale (twice the weight of the other items). For all of these items, 0 is the "best" rating and the highest score (2 or 4) is the "worst" rating. The sum of the scores from the first 17 items; 0-7 =Normal; 8-13 =mild depression; 14-18 =moderate depression; 19-22 =severe depression; ≥23 =very severe depression. The total score ranges from 0 to 52, with higher score indicating worse depressive symptoms.
Time Frame: Baseline and Week 14
Population: Efficacy Sample comprised all participants in Safety Sample who had end of Phase A value and at least one post-randomization efficacy evaluation for MADRS total score in Phase B. The Last-observation-carried-forward (LOCF) data set included data recorded at Phase B visit, if no observation was recorded, data was carried forward from previous visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 183 | 188
Units on a scale | -5.89 (0.48) | -3.55 (0.47)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; ANCOVA_Last observation carry forward (LOCF) model with treatment and trial site as main effects, and baseline (end of Phase A [Week 8]) value as a covariate was used; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -2.34, 95% CI 2-sided [-3.47 to -1.22]

16. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) to Week 14 in HAM-D Rating Scale Total Score for the Efficacy Sample Per the Final Protocol.
Description: as for outcome 15
Time Frame: Baseline and Week 14
Population: All participants in the efficacy sample who met the revised randomization criteria for incomplete response as defined in protocol amendment 3. The LOCF data set included data recorded at Phase B visit, if no observation was recorded, data was carried forward from previous visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 172 | 175
Units on a scale | -5.89 (0.51) | -3.59 (0.49)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Test type: Superiority or Other; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -2.29, 95% CI 2-sided [-3.47 to -1.12]

17. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) to Week 14 in Hamilton Anxiety (HAM-A) Rating Scale Total Score for the Efficacy Sample
Description: The HAM-A is utilized for the evaluation of anxiety symptoms. The HAM-A consists of 14 items. Each item is rated on a 0 to 4 scale. For all of these items, 0 is the "best" rating and 4 is the "worst" rating. If no item scores are missing, then the HAM-A total score is the sum of all 14 item scores. The possible total scores are from 0 to 56, with higher scores indicating worse anxiety symptoms.
Time Frame: Baseline and Week 14
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 181 | 188
Units on a scale | -3.94 (0.43) | -2.77 (0.42)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; ANCOVA_LOCF model with treatment and trial site as main effects, and baseline (end of Phase A [Week 8]) value as a covariate was used; Test type: Superiority or Other; p = 0.0219, ANCOVA; Mean Difference (Final Values) = -1.17, 95% CI 2-sided [-2.17 to -0.17]

18. Secondary Outcome: Change From Baseline (End of Phase A [Week 8]) to Week 14 in HAM-A Rating Scale Total Score for the Efficacy Sample Per the Final Protocol.
Description: as for outcome 17
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 171 | 175
Units on a scale | -3.79 (0.45) | -2.70 (0.43)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Test type: Superiority or Other; p = 0.0376, ANCOVA; Mean Difference (Final Values) = -1.09, 95% CI 2-sided [-2.13 to -0.06]

19. Secondary Outcome: Percentage of Participants With MADRS Response at Week 14 Relative to Baseline (End of Phase A [Week 8]) for the Efficacy Sample.
Description: The MADRS response was defined as >/=50% reduction in MADRS total score from end of Phase A (Week 8).
Time Frame: Baseline and Week 14
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 187 | 191
Percentage of participants | 23.5 | 14.7
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Test type: Superiority or Other; p = 0.0176, Cochran-Mantel-Haenszel; CHM general association test controlling for trial site; Ratio of Response Rate = 1.63, 95% CI 2-sided [1.09 to 2.44]

20. Secondary Outcome: Percentage of Participants With MADRS Response at Week 14 Relative to Baseline (End of Phase A [Week 8]) for the Efficacy Sample Per the Final Protocol.
Description: The MADRS response was defined as >/=50% reduction in MADRS total score from end of Phase A (Week 8).
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 175 | 178
Percentage of participants | 23.4 | 15.7
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Test type: Superiority or Other; p = 0.0429, Cochran-Mantel-Haenszel; CHM general association test controlling for trial site; Ratio of Response Rate = 1.54, 95% CI 2-sided [1.01 to 2.35]

21. Secondary Outcome: Percentage of Participants With MADRS Remission at Week 14 Relative to Baseline (End of Phase A [Week 8]) for the Efficacy Sample.
Description: MADRS remission was defined as </=10 and >/=50% reduction in MADRS total score from end of Phase A (Week 8).
Time Frame: Baseline and Week 14
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 187 | 191
Percentage of participants | 14.4 | 8.38
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Test type: Superiority or Other; p = 0.0586, Cochran-Mantel-Haenszel; CHM general association test controlling for trial site; Ratio of Remission Rate = 1.68, 95% CI 2-sided [0.98 to 2.86]

22. Secondary Outcome: Percentage of Participants With MADRS Remission at Week 14 Relative to Baseline (End of Phase A [Week 8]) for the Efficacy Sample Per the Final Protocol.
Description: MADRS remission was defined as </=10 and >/=50% reduction in MADRS total score from end of Phase A (Week 8).
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 175 | 178
Percentage of participants | 14.9 | 8.99
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Test type: Superiority or Other; p = 0.0671, Cochran-Mantel-Haenszel; CHM general association test controlling for trial site; Ratio of Remission Rate = 1.67, 95% CI 2-sided [0.97 to 2.90]

23. Secondary Outcome: Percentage of Participants With CGI-I Scale Response Rate at Week 14 Relative to Baseline (End of Phase A [Week 8]) for the Efficacy Sample.
Description: CGI-I response was defined as a CGI-I score of 1 (very much improved) or 2 (much improved).
Time Frame: Baseline and Week 14
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 187 | 191
Percentage of participants | 44.4 | 27.7
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel; CHM general association test controlling for trial site; Ratio of Response Rate = 1.61, 95% CI 2-sided [1.23 to 2.10]

24. Secondary Outcome: Percentage of Participants With CGI-I Scale Response Rate at Week 14 Relative to Baseline (End of Phase A [Week 8]) for the Efficacy Sample Per the Final Protocol.
Description: CGI-I response was defined as a CGI-I score of 1 (very much improved) or 2 (much improved).
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Number; unit: Percentage of participants
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Number analyzed (Participants) | 175 | 178
Percentage of participants | 43.4 | 26.4
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg/Day + ADT vs Double-blind Placebo + ADT; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; CHM general association test controlling for trial site; Ratio of Response Rate = 1.69, 95% CI 2-sided [1.27 to 2.27]

ADVERSE EVENTS:
Time Frame: Adverse Events with an onset date on or after the start of double-blind treatment and occurring up to 30 days after the last day of double-blind treatment were included.
Description: Safety sample comprised of randomized participants in Phase B who received at least one dose of double-blind trial medication. Participants were excluded only if there was evidence that the participant did not take trial medication. If a participant was dispensed trial medication and is lost to follow-up that participant was considered exposed.
Arm/Group | Brexpiprazole 2 mg/Day + ADT | Double-blind Placebo + ADT
Serious Adverse Events (participants affected / at risk) | 2/188 | 2/191
Other Adverse Events (participants affected / at risk) | 37/188 | 27/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 2 mg/Day + ADT (N=188) | Double-blind Placebo + ADT (N=191)
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Comminuted Fracture (Injury, poisoning and procedural complications) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 2 mg/Day + ADT (N=188) | Double-blind Placebo + ADT (N=191)
Diarrhoea (Gastrointestinal disorders) | 5 | 10
Upper resporatory tract infection (Infections and infestations) | 6 | 12
Weight increased (Investigations) | 15 | 6
Akathisia (Nervous system disorders) | 14 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No